CLINICAL TRIAL: NCT04830436
Title: Analysis of the Impact of Undernutrition in Patients Over 70 Years of Age Thrombolysed and/or Thrombectomized for Stroke
Brief Title: Impact of Undernutrition in Patients Over 70 Years of Age Thrombolysed and/or Thrombectomized for Stroke
Acronym: Denut_AVC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Denutrition_AVC2
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Undernutrition is a frequent problem in hospitals (at least 30% of patients, SENECA-NHANES studies). Its impact on morbidity and mortality is well known in gerontology, oncology and intensive care. There are very few neurovascular studies dealing with the consequences of undernutrition present before the stroke. Indeed, most of the medical literature concerns only undernutrition acquired after a stroke. The investigator propose to analyze medical data from a cohort of patients over 70 years of age thrombolysed and/or thrombectomized in the neurovascular department between the years 2014 and 2019.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years of age with cerebral infarction, thrombolysed and/or thrombectomized between 2014 and 2019, managed in the Neurology and Neurovascular Department of the Paris Saint-Joseph Hospital
* French-speaking patient

Exclusion Criteria:

* Patients with non-thrombolyzed stroke
* Patient with a TIA (Transient Ischemic Attack)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patients who object to the use of their data for this research

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized for cerebral infarction who received thrombolysis and/or thrombectomy treatment between 2014 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution of the patients: NIHSS | Day 5
  This outcome correspond to the National Institute of Health Stroke Score (NIHSS) at day 5. The score is 0: No stroke symptoms; 1-4: Minor stroke; 5-15: Moderate stroke; 16-20: Moderate to severe stroke; 21-42 : Severe stroke.
Modified Rankin Scale | Month 3
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Rankin scale: 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruandet, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Zhang J, Zhao X, Wang A, Zhou Y, Yang B, Wei N, Yu D, Lu J, Chen S, Wang Y, Wang C, Xue R, Zhang Y, Li Y, Yu L, Wang S, Chen Z, Zheng T, Zhang Z, Xia M, He M, Li W, Zhang Z, Zeng F, Chen S, Fu Y, Liu G, Wang L, Huang Z, Ma J, Mu F, Xu Y, Huang R, Wang L, Wang Y. Emerging malnutrition during hospitalisation independently predicts poor 3-month outcomes after acute stroke: data from a Chinese cohort. Asia Pac J Clin Nutr. 2015;24(3):379-86. doi: 10.6133/apjcn.2015.24.3.13. PMID 26420177
- [Background] Yoo SH, Kim JS, Kwon SU, Yun SC, Koh JY, Kang DW. Undernutrition as a predictor of poor clinical outcomes in acute ischemic stroke patients. Arch Neurol. 2008 Jan;65(1):39-43. doi: 10.1001/archneurol.2007.12. PMID 18195138
- [Background] Unosson M, Ek AC, Bjurulf P, von Schenck H, Larsson J. Feeding dependence and nutritional status after acute stroke. Stroke. 1994 Feb;25(2):366-71. doi: 10.1161/01.str.25.2.366. PMID 8303747
- [Background] Euronut - SENECA. Nutrition and the elderly in Europe. 1st European Congress on Nutrition and Health in the Elderly. The Netherlands, December 1991. Eur J Clin Nutr. 1991 Dec;45 Suppl 3:1-196. No abstract available. PMID 1687315